CLINICAL TRIAL: NCT00697138
Title: Agonist Replacement Therapy for Cocaine Dependence: Identifying Novel Medications
Brief Title: Agonist Replacement Therapy for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Princpal Investigator, University of Kentucky
Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DA021155; Agonists for Cocaine Abuse; R01DA021155 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Dependence; Pharmacotherapies
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: d-Amphetamine; Atomoxetine

INTERVENTIONS:
Drug: d-Amphetamine; Atomoxetine — Dexedrine (0-60 mg/day); Strattera (0-80 mg/day)

SUMMARY:
Cocaine dependence is a significant public health concern. The proposed research will provide important clinical information regarding the efficacy of agonists replacement therapies for managing cocaine dependence.

DETAILED DESCRIPTION:
Cocaine abuse and dependence continue to be significant public health concerns. The number of Americans that used cocaine in the past month, the percentage of 12th-, 10th- and 8th-graders that used cocaine in the past year, and the percentage of treatment admissions involving cocaine has remained stable in recent years. In 1996, cocaine use cost society over $45 billion due to medical consequences, lost productivity and crime. Because of the public-health concerns and costs associated with its abuse, identifying a pharmacotherapy for cocaine dependence is a priority with the National Institute on Drug Abuse (N.I.D.A.). A pharmacological adjunct for cocaine dependence has not yet been identified.

The results of clinical trials suggest that agonist replacement therapies (e.g., d-amphetamine) may be effective for cocaine dependence. Because d-amphetamine reduces cocaine use, these clinical findings can be used as a reference to identify human laboratory procedures for screening putative pharmacotherapies. Identifying procedures for assessing the efficacy of putative pharmacotherapies is important because human laboratory studies can be conducted more rapidly and efficiently than clinical trials. The present project has two specific aims. The first specific aim is to demonstrate the sensitivity and predictive validity of human laboratory procedures commonly used to screen putative pharmacotherapies for cocaine dependence. To accomplish this aim, we will conduct two "proof-of-concept" studies. We will first demonstrate the safety and tolerability of d-amphetamine-cocaine combinations (Exp. 1). We will then demonstrate that d-amphetamine maintenance attenuates the reinforcing effects of cocaine (Exp. 2). The ability to attenuate the reinforcing effects of cocaine may be an important characteristic of an effective pharmacotherapy. The results of these studies will help elucidate the optimal conditions (e.g., dose) under which d-amphetamine might be expected to be effective. The second specific aim is to determine the efficacy of atomoxetine (Strattera®) as a putative agonist replacement pharmacotherapy for cocaine dependence. To accomplish this aim, we will conduct two experiments to determine the effects of cocaine during atomoxetine maintenance. We will first demonstrate the safety and tolerability of atomoxetine-cocaine combinations (Exp. 3). Finally, we will determine the reinforcing effects of intranasal cocaine during atomoxetine maintenance (Exp. 4). Atomoxetine, a potent norepinephrine uptake blocker, was chosen for study because its pharmacological and behavioral effects overlap to some extent with those of d-amphetamine, but it appears to have less abuse potential. Identifying novel agonist replacement therapies is important because clinicians may be reluctant to use d-amphetamine because of its abuse potential.

ELIGIBILITY:
Inclusion Criteria:

Must meet diagnostic criteria for cocaine dependence Current cocaine use at study entry, as determined by urine screen Body Mass Index less or equal to 30 ECG results within normal limits If female, willing to use contraception throughout study

Exclusion Criteria:

Meets diagnostic criteria for dependence on drug other than cocaine and nicotine Currently seeking treatment for substance abuse Current or past history of serious illness including impaired heart function, seizures and central nervous system tumors Family history o heart disease or seizures Current of past psychiatric disorder other than substance abuse Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2006-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Behavioral effects of cocaine | Measure throughout the study

SECONDARY OUTCOMES:
Heart rate; blood pressure; ECG | Measure throughtout study

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Rush, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States